CLINICAL TRIAL: NCT02453139
Title: Evasion of Immune Editing by Circulating Tumour Cells in an Exercise Modifiable Mechanism Underlying Aggressive Behaviour in Obese Men With Prostate Cancer
Brief Title: Exercise, Prostate Cancer and Circulating Tumour Cells
Acronym: ExPeCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Prof Stephen Finn, Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202370
Record Dates: First submitted 2015-05-12; First posted 2015-05-25 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer; Obesity
MeSH Terms: conditions — Prostatic Neoplasms; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise group (Experimental): 6 month supervised and home based moderate intensity aerobic exercise programme
  Interventions: Behavioral: Exercise
- Control (No Intervention): Non-exercising control group receiving usual care

INTERVENTIONS:
Behavioral: Exercise — 6 month supervised and home based aerobic exercise intervention
  Arms: Exercise group

SUMMARY:
Obesity, known to be associated with a pro-inflammatory, pro-thrombotic humoral milieu, confers a worse prognosis in prostate cancer (PrCa). Circulating tumour cells (CTCs) are identified in the blood in advanced cancer. Their quantitation provides prognostic information. "Cloaking" of CTCs by adherent platelets impedes natural killer (NK)-cell clearance of CTCs from the circulation, enhancing metastatic spread. NK-cell function in blood and in solid organs is quantitatively and qualitatively reduced in obesity. Platelet cloaking may be enhanced in obesity due to the pro-inflammatory, pro-thrombotic state, and may be a mechanism for worse cancer-specific outcomes in this group. Obesity and its biochemical effects may be influenced by lifestyle changes such as exercise. Physical activity reduces levels of systemic inflammatory mediators and so an aerobic exercise intervention may represent an accessible and cost-effective means of ameliorating the pro-inflammatory effects of obesity. The ExPeCT trial will determine if a prescribed exercise intervention can ameliorate the degree of platelet cloaking in obese and non-obese men with advanced prostate cancer.

DETAILED DESCRIPTION:
The overarching hypothesis is that enhanced platelet cloaking of circulating tumour cells in obese men with prostate cancer, due to increased systemic inflammation, is a mechanism underlying worse prognosis of cancer in these patients.

The investigators aim to test the following four hypotheses, dividing the experimental and analytical work into four separate projects.

1. Platelet cloaking of circulating PrCa tumour cells is more prominent in men with obesity than without
2. Regular exercise can ameliorate platelet cloaking
3. The degree of platelet cloaking varies with levels of systemic and primary tumour inflammation and coagulability
4. Expression of an obesity-associated lethality gene signature leads to variation in platelet cloaking

For the first hypothesis, 200 men with metastatic PrCa will be recruited, and divided into exposed and non-exposed groups based on body mass index (BMI >25). The objective will be to enumerate CTCs and quantify the degree of platelet cloaking in exposed and non-exposed groups, and to draw meaningful comparisons between the two.

For the second hypothesis, the objective will be to determine to what extent the number of CTCs and the degree of platelet cloaking varies in exposed and non-exposed groups following a supervised exercise intervention, and to compare this with a non-exercised comparison group. The exercise intervention will prescribe moderate intensity aerobic exercise that will be supervised once per week for 3 months and completed independently at home for a further 3 months. Patients will wear Polar heart rate monitors to monitor exercise prescription and progression. Assessments including blood sampling and quality of life questionnaires will be completed at baseline, 3 months and 6 months.

For the third hypothesis, the objective will be to build a serological, haematological and immunological picture of the state of systemic inflammation and coagulability, and the degree of inflammation within the prostate gland. Furthermore, the investigators intend to correlate and compare these variables with the results of the first and second objectives, in order to determine whether the number of CTCs and the degree of platelet cloaking varies with changes in the inflammatory / coagulatory milieu.

For the fourth hypothesis, the objective will be to determine whether the expression profile of a number of lethality-associated genes, known to be associated with PrCa progression, coagulation and stem-cell like phenotype, correlates with the number of CTCs and the degree of their cloaking by platelets.

CTC numbers and the degree of platelet cloaking will be common denominators which anchor these four objectives together and enable comparison between them.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before any study-related procedures
2. Age ≥ 18 years and male
3. Histologically confirmed diagnosis of prostate adenocarcinoma
4. Metastatic disease as confirmed by CT/MRI or by bone scan
5. Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections, or major surgery within 28 days prior to randomisation
6. Capable of participating safely in the proposed exercise intervention as assessed and signed off by a treating physician involved in ExPeCT recruitment.

Exclusion Criteria:

1. No history of radical prostatectomy
2. No previous diagnosis of any other malignant tumour (patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded provided they have undergone complete resection)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in Platelet cloaking of Circulating Tumour Cells | Change from baseline in platelet cloaking of circulating tumours cells at 3 months and 6 months
  Enumeration of circulating tumour cells and degree of platelet cloaking of CTCs

SECONDARY OUTCOMES:
Change in systemic inflammation | Change in cytokines from baseline in inflammation at 3 months and 6 months
  Blood samples will be taken from participants at each assessment and analysed by multi-plex assays for levels of cytokines (TNF-alpha and interleukin (IL)-6
Change in Quality of Life Questionnaire | Change from baseline in quality of life at 3 months and 6 months
  Participants will complete quality of life questionnaires assessing a range of issues including sleep, diet quality and physical activity at each assessment

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Finn, Principal Investigator — University of Dublin, Trinity College
Locations (6):
- Ireland (5):
  - Adelaide and Meath Incorporating the National Children's Hospital, Tallaght, Dublin
  - St James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St Luke's Hospital, Dublin
- Guy's St Thomas, London, United Kingdom

REFERENCES:
- [Derived] Sheill G, Brady L, Hayes B, Baird AM, Guinan E, Vishwakarma R, Brophy C, Vlajnic T, Casey O, Murphy V, Greene J, Allott E, Hussey J, Cahill F, Van Hemelrijck M, Peat N, Mucci L, Cunningham M, Grogan L, Lynch T, Manecksha RP, McCaffrey J, O'Donnell D, Sheils O, O'Leary J, Rudman S, McDermott R, Finn S. ExPeCT: a randomised trial examining the impact of exercise on quality of life in men with metastatic prostate cancer. Support Care Cancer. 2023 Apr 22;31(5):292. doi: 10.1007/s00520-023-07740-4. PMID 37086362
- [Derived] Brady L, Hayes B, Sheill G, Baird AM, Guinan E, Stanfill B, Vlajnic T, Casey O, Murphy V, Greene J, Allott EH, Hussey J, Cahill F, Van Hemelrijck M, Peat N, Mucci L, Cunningham M, Grogan L, Lynch T, Manecksha RP, McCaffrey J, O'Donnell D, Sheils O, O'Leary J, Rudman S, McDermott R, Finn S. Platelet cloaking of circulating tumour cells in patients with metastatic prostate cancer: Results from ExPeCT, a randomised controlled trial. PLoS One. 2020 Dec 18;15(12):e0243928. doi: 10.1371/journal.pone.0243928. eCollection 2020. PMID 33338056
- [Derived] Sheill G, Guinan E, Neill LO, Hevey D, Hussey J. The views of patients with metastatic prostate cancer towards physical activity: a qualitative exploration. Support Care Cancer. 2018 Jun;26(6):1747-1754. doi: 10.1007/s00520-017-4008-x. Epub 2017 Dec 14. PMID 29243168
- [Derived] Sheill G, Brady L, Guinan E, Hayes B, Casey O, Greene J, Vlajnic T, Cahill F, Van Hemelrijck M, Peat N, Rudman S, Hussey J, Cunningham M, Grogan L, Lynch T, Manecksha RP, McCaffrey J, Mucci L, Sheils O, O'Leary J, O'Donnell DM, McDermott R, Finn S. The ExPeCT (Examining Exercise, Prostate Cancer and Circulating Tumour Cells) trial: study protocol for a randomised controlled trial. Trials. 2017 Oct 4;18(1):456. doi: 10.1186/s13063-017-2201-3. PMID 28978344